CLINICAL TRIAL: NCT02197559
Title: A Prospectie Cohort Study of Bare -Metal Stents and Drug -Eluting Stents in the Treatment of Patients With Vertebral Artery Ostium Stenosis
Brief Title: Bare -Metal Stents and Drug -Eluting Stents in the Treatment of Patients With Vertebral Artery Ostium Stenosis
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: BEST-VAOS
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2014-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke, restenosis,bare-metal stents, drug -eluting stents
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BMS group, DES group: All the participants in this group will be performed with bare-metal stents or drug -eluting stents
  Interventions: Procedure: DES group; Procedure: BMS group

INTERVENTIONS:
Procedure: DES group — all the participants in this group will be performed with drug -eluting stents
  Other Names: Drug -eluting stents group
Procedure: BMS group — all the participants in this group will be performed with bare-metal stents
  Other Names: Bare-metal stents group

SUMMARY:
The study hypothesizes that Drug -eluting stents are more effective in preventing restenosis than Bare-metal stents after Vertebral Artery Ostium stenting

DETAILED DESCRIPTION:
The vertebral artery ostium stenosis was one of the higher risk of the ischemia stroke in China. In the mean time ,more and more people accept revascularization. There are no prospective studies for comparison of prevention of restenosis after Drug -eluting stents and Bare-metal stents until now.

The main aim of this study is to observe the following details:

1. Late loss in lumen diameter in follow-up ≥50%
2. Death, non -fatal stroke 30 days after stent implantation associated with antiplatelet drugs
3. Death, non -fatal stroke 12 months after stent implantation associated with antiplatelet drugs

Secondary endpoint:

brain, gastrointestinal and urinary system bleeding in 12 months follow-up

ELIGIBILITY:
Inclusion Criteria:

- symptomatic posterior circulation ischemia including monor stroke (mRS ≤2) or TIA result from the stenosis in the vertebral artery ostium.

70% to 99% stenosis of vertebral artery ostium.

Exclusion Criteria:

* etiology of stenotic lesions not atherosclerosis patients had undergone previos interventions on the vertebral artery ostium ipsilateral severe stenotic lesions in subclavian artery involved as well as vertebral artery ostium

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic status: as evidenced by TIA or non-severe stroke within the past 12 months attributed to 70% to 99% stenosis of vertebral artery ostium are eligible. Degree of stenosis: >70% and <99%; stenosis may be diagnosed by TCD, MRA, or CTA to qualify for angiogram performed as part of the study protocol, but must be confirmed by catheter angiography for enrollment in the trial. All the patients should be performed with PTAS beyond a duration of 3 weeks from the latest ischemic symptom onset. No fresh infarctions identified on MRI (indicated as high signals on DWI series) upon enrollment.Patient is willing and able to return for all follow-up visits required by the protocol Patient understands the purpose and requirements of the study, can make him/herself understood, and has signed informed consent.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Late loss in lumen diameter in follow-up ≥50% | 1 year
  Late loss in lumen diameter in follow-up ≥50%
Death, non -fatal stroke 30 days after stent implantation associated with antiplatelet drugs | 30 days
  Death, non -fatal stroke 30 days after stent implantation associated with antiplatelet drugs
Death, non -fatal stroke 12 months after stent implantation associated with antiplatelet drugs | 12 months
  Death, non -fatal stroke 12 months after stent implantation associated with antiplatelet drugs

SECONDARY OUTCOMES:
brain, gastrointestinal and urinary system bleeding in 12 months follow-up | 12 months
  brain, gastrointestinal and urinary system bleeding in 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ling, M.D., Principal Investigator — Xuanwu Hospital, Capital University of Medical Sciences, Beijing, China
Locations (1):
- Department of neurosurgery, Xuanwu hospital, Beijing, China